CLINICAL TRIAL: NCT05411380
Title: Tucidinostat Combined With Metronomic Capecitabine and Endocrine Therapy for Advanced HR-positive, HER2-negative Breast Cancer After CDK4/6 Inhibitor：a Prospective, Single-arm, Phase II Clinical Trial.
Brief Title: Tucidinostat Combined With Metronomic Capecitabine and Endocrine Therapy for Advanced HR-positive, HER2-negative Breast Cancer After CDK4/6 Inhibitor.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: wang shusen (Other)
Responsible Party: Sponsor-Investigator, wang shusen, Chief Physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-020
Record Dates: First submitted 2022-06-05; First posted 2022-06-09 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: metronomic capecitabine; endocrine therapy; histone deacetylase inhibitor; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Capecitabine; Anastrozole; Letrozole; exemestane; Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tucidinostat+Metronomic Capecitabine+Endocrine Therapy (Experimental): This arm is divided into two groups. The main difference of this two groups lies in the selection of endocrine therapy. One is supposed to choose aromatase inhibitor, and the other is fulvestrant. The principle of making choice is based on the history of endocrine drug use.
  Interventions: Drug: Tucidinostat; Drug: Capecitabine; Drug: Endocrine Therapy

INTERVENTIONS:
Drug: Tucidinostat — 20mg each time, orally 30 minutes after dinner, 3 weeks for a cycle, administered on day 1, day 4, day 8, day 11, day 15,and day 18 of each cycle (twice a week, at least 3 days between each administration)
  Other Names: Chidamide
Drug: Capecitabine — 500mg orally three times a day (continuously)
  Other Names: Xeloda
Drug: Endocrine Therapy — Anastrozole, 1mg, orally once daily or Letrozole, 2.5mg, orally once daily or Exemestane , 25mg, orally once daily or fulvestrant 500 mg each time, intramuscularly, injected on the 1st day and 15th day of the 1st cycle, and on the 1st day for subsequent cycle( 4 weeks for one cycle)
  Other Names: Anastrozole; Letrozole; Exemestane; Fulvestrant

SUMMARY:
The study is designed to explore the clinical benefit following treatment with tucidinosta in combination with metronomic capecitabine and endocrine therapy in patients with hormone receptor-positive, Her2-negative advanced breast cancer who have received CDK4/6 Inhibitor treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, and ≤75 years old, female; 2. Histologically confirmed HR positive and HER2 negative postmenopausal metastatic breast cancer patients [HER2 negative is defined as immunohistochemistry(IHC) 0 or IHC 1+, and if the score of IHC is 2+, fluorescence in situ hybridization technology (FISH) test must be negative, HR positve is defined as ER or PR ≥1%;]; 3. After the failure of previous CDK4/6 inhibitor therapy; 4.Receive one line of chemotherapy at most; 5.Premenopausal women need to take effective measures to suppress ovarian function, such as drug suppression, oophorectomy; 6.ECOG score 0-1; 7. According to RECIST1.1 criteria, at least there is one measurable lesion or simple bone metastasis; 8. The main organ and bone marrow function levels meet the following requirements:

1. Blood routine: neutrophil (ANC) ≥ 1.5×109/L; platelet count (PLT) ≥ 90× 109/L; hemoglobin (Hb) ≥ 90g/L; It is required that no blood products (including red blood cells and platelet products, etc.) have been transfused and no growth factors (including colony-stimulating factor, interleukin, and erythropoietin, etc.) have been used for supportive treatment within 2 weeks before the examination.
2. Liver function: serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (with liver Requirements for metastatic patients: ALT and AST≤5×ULN);
3. Renal function: serum creatinine (Cr)≤1.5×ULN or creatinine clearance rate>60mL/min;

9. Expected survival time ≥ 3 months; 10. Voluntary participation study, signed written informed consent.

Exclusion Criteria:

1. Known hypersensitivity to any formulation component of the study drug;
2. patients with previous severe, unexpected reactions to fluoropyrimidines or known hypersensitivity to fluoropyrimidines;
3. Patients with complete deficiency of dihydropyrimidine dehydrogenase (DPD) activity;
4. Visceral crisis;
5. Previously received treatment with histone deacetylase inhibitors or fluoropyrimidine drugs such as capecitabine;
6. Received chemotherapy, targeted therapy, Chinese herbal medicine with anti-tumor indications, or immunomodulatory drugs (including thymosin, interferon, interleukin, etc.) within 4 weeks before enrollment, or still within 5 half-lives of such drugs;
7. Received palliative radiotherapy for local lesions within 4 weeks before enrollment;
8. Patients with gastrointestinal perforation, fistula, abdominal abscess, gastrointestinal ulcer or active diverticulosis before enrollment;
9. Significant malnutrition (weight loss > 5% in the past 1 month or > 15% in the past 3 months, or food intake decreased by 1/2 or more in the past week), or still need to rely on intravenous nutritional support during the screening period;
10. Toxicities that did not recover to National Cancer Institute Common Adverse Event Terminology Version 5.0 (NCICTCAEv5.0) grade 0 or 1 toxicity from prior antineoplastic therapy prior to the first dose of study treatment(alopecia, grade 2 fatigue, grade 2 anemia, non-clinically critical and asymptomatic laboratory abnormalities can be enrolled);
11. Patients with currently symptomatic brain or meningeal metastasis;
12. Received immunosuppressive drugs within 4 weeks before enrollment, excluding nasal spray, inhalation or other local glucocorticoids or physiological doses systemic glucocorticoids (no more than 10 mg/day of prednisone or other glucocorticoids at an equivalent dose), or use of glucocorticoids for the prevention of contrast medium allergy;
13. The patient has any active autoimmune disease or has history of immune disorders (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism; patients with vitiligo or complete remission of asthma in childhood without any intervention in adulthood can be included; those with asthma that require medical intervention with bronchodilators are not included);
14. Patients with active pulmonary tuberculosis who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before screening;
15. Complications requiring long-term use of immunosuppressive drugs, or systemic or topical use of corticosteroids with immunosuppressive doses;
16. Received any anti-infection vaccine (such as influenza vaccine, chickenpox vaccine, etc.) within 4 weeks before enrollment;
17. Received major surgery (craniotomy, thoracotomy or laparotomy) within 4 weeks before enrollment or is expected to undergo major surgery during the study treatment period; received exploratory laparoscopic surgery within 2 weeks prior to enrollment;received central venous catheterization within 7 days prior to enrollment;
18. Concurrent participation in another interventional clinical study, unless participating in an observational (non-interventional) clinical study or in the safety follow-up of an interventional study Stage;
19. Known acute or chronic active hepatitis B (HBsAg positive and HBV DNA virus Load ≥ULN or ≥10^3 copies/mL) or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive);
20. Severe heart disease or discomfort, including but not limited to the following diseases: 1) Diagnosed history of heart failure or systolic dysfunction (LVEF<50%); 2) arrhythmias requiring medical treatment or clinically significant; 3) high-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate > 100 bpm, significant ventricular arrhythmia (such as ventricular tachycardia) or higher-grade AV block (ie Mobitz II second-degree AV block or third-degree AV block); 4) Angina pectoris; 5 ) Clinically significant valvular heart disease; 6) ECG shows transmural myocardial infarction; 7) Any other heart disease judged by the investigator to be inappropriate to participate in this trial, etc.;
21. Inability to swallow, bowel obstruction, or other factors that interfere with drug taking and absorption;
22. A history of immunodeficiency, including HIV test positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
23. Pregnant, lactating female patients, female patients of childbearing potential with a positive baseline pregnancy test, or patients of childbearing age who are unwilling to use effective contraception throughout the trial and within 6 months after the last study drug;
24. Serious concomitant disease or other comorbidities that would interfere with planned treatment;
25. Any other conditions deemed inappropriate by the investigator to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 3 years
  Objective response is defined as a complete response (CR) or partial response (PR) according to RECIST v.1.1 recorded from randomization until disease progression or death due to any cause

SECONDARY OUTCOMES:
Progress-free survival | Up to 3 years
  Time from randomization to the first documentation of objective tumor progression or to death due to any cause.
Disease Control Rate | Up to 3 years
  Disease control is defined as complete response (CR), partial response (PR), or stable disease (SD) ≥24 weeks according to the RECIST version 1.1 recorded in the time period between randomization and disease progression or death to any cause.
Overall Survival | Up to 3 years
  Time from randomization to date of death due to any cause. according to the RECIST version 1.1 recorded in the time period between randomization and disease progression or death to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Susen Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Shusen Wang, Guangzhou, Gangdong, China

IPD SHARING:
Plan to Share IPD: Undecided